CLINICAL TRIAL: NCT02755935
Title: Implantation With the Cochlear Nucleus® CI532 Implant - Early Experience Study
Brief Title: CI532 - Early Experience Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5660
Record Dates: First submitted 2016-04-19; First posted 2016-04-29 (Estimated); Results first posted 2018-02-22 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-01

CONDITIONS: Sensorineural Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implanted (Experimental): Subjects who meet the specified inclusion criteria and are implanted with the CI532 cochlear implant
  Interventions: Device: Cochlear Nucleus CI532

INTERVENTIONS:
Device: Cochlear Nucleus CI532 — cochlear implantation

SUMMARY:
To evaluate performance outcomes in patients implanted with the Cochlear Nucleus CI532 electrode array.

DETAILED DESCRIPTION:
To compare speech perception and audiometric outcomes in patients implanted with the Cochlear Nucleus CI532 electrode array at 3 months postactivation with their best preoperative hearing status.

ELIGIBILITY:
Inclusion Criteria:

* Medical and audiological candidate for a CI532 cochlear implant per commercially approved, age appropriate, FDA indications
* Post-linguistically deafened
* Ability to complete age appropriate testing

Exclusion Criteria:

* Previous cochlear implantation in the ear to be implanted
* Pre-linguistically deafened (onset of hearing loss at less than two years of age)
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array
* Diagnosis of retro-cochlear pathology
* Diagnosis of auditory neuropathy
* Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure and use of the prosthetic device
* Unwillingness or inability to comply with all investigational requirements
* Additional cognitive handicaps that would prevent participation on all study requirements

Min Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - NorthShore University, Skokie, Illinois
  - University of Iowa, Iowa City, Iowa
  - The University of Michigan, Ann Arbor, Michigan
  - Center for Hearing and Balance, Chesterfield, Missouri
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dallas Ear Institute, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Implanted
Started | 24
Completed | 22
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Implanted
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Speech understanding (% correct) on AzBio sentences in quiet in the ear to be implanted [Mean (Standard Deviation); unit: percent correct] | 11.2 (16.6)
Speech understanding (% correct) on AzBio sentences in noise in the ear to be implanted [Mean (Standard Deviation); unit: percent correct] | 5.3 (12.8)

OUTCOME MEASURES:

1. Primary Outcome: Speech Understanding (% Correct) on AzBio Sentences in Quiet in the Implanted Ear
Description: Unilateral listening performance at 3 months post activation with the CI532 compared to the best aided unilateral preoperative condition for sentence perception in quiet.
Time Frame: 3 months postactivation of the sound processor
Population: implanted and enrolled
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Implanted
Number analyzed (Participants) | 22
percent correct | 53.5 (28.2)

2. Primary Outcome: Speech Understanding (% Correct) on AzBio Sentences in Noise in the Implanted Ear
Description: unilateral listening performance at 3 months post activation with the CI532 compared to the best aided unilateral preoperative condition for sentence perception in noise
Time Frame: 3 months post-activation
Population: implanted and enrolled
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Implanted
Number analyzed (Participants) | 22
percent correct | 25.3 (24.5)

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Implanted
All-Cause Mortality (participants affected / at risk) | 1/24
Serious Adverse Events (participants affected / at risk) | 2/24
Other Adverse Events (participants affected / at risk) | 6/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted (N=24)
death (General disorders) | 1 (1) — death from recurrence of a previous medical condition unrelated to the device or procedure
skin flap (Infections and infestations) | 1 (1) — Incision breakdown, revised successfully in the OR
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implanted (N=24)
Facial nerve (Ear and labyrinth disorders) | 1 (1) — Facial nerve weakness following surgery, Treated with oral medications and resolved.
Vertigo or dizziness (Ear and labyrinth disorders) | 1 (1) — with stimulation of specific electrodes
Tingling sensation (Ear and labyrinth disorders) | 1 (1) — tingling/shocking with stimulation of specific electrodes. Programmed around, resolved
Device related/programming problems (Product Issues) | 3 (3) — open circuit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT02755935/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT02755935/SAP_001.pdf